CLINICAL TRIAL: NCT00586222
Title: Neurometabolic Effects of the Essential Polyunsaturated Fatty Acids in Early-Onset Bipolar Disorder: A Magnetic Resonance Spectroscopy Study
Brief Title: Omega 3 Fatty Acid Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sencan Solay Unal, M.D. P, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 06-004285
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Omega-3 Fatty Acids; Pediatric Bipolar Disorder; Adolescent Bipolar Disorder; Magnetic Resonance Spectroscopy Imaging
Keywords: Omega-3 Fatty Acids; Pediatric Bipolar Disorder; Adolescent Bipolar Disorder; MRS
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Placebo Comparator)
  Interventions: Other: Placebo
- Healthy Comparsions (No Intervention): We will compare the BP group with 32 age-, gender-, and handedness-matched healthy adolescents. Subjects who have a first or second degree relative with a psychiatric history will be excluded from the healthy comparison group. Subjects must be safe to undergo MRI scanning as per Mayo MRI safety screening which is explained in detail elsewhere in this protocol. We will exclude the subjects with cardiac pacemakers, metallic clips, other bodily metallic implants and dental braces because of the MRS procedure. Subjects who cannot complete clinical assessments or the MRI scan and subjects who are not fluent in English will be excluded from the study.
- 1 (Experimental)
  Interventions: Dietary Supplement: Omega-3 Fatty Acid

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid — 600 mg of eicosapentaenoic acid, 340 g of docosahexanoic acid, and 96 mg gama-linoleic acid for 12 weeks.
  Arms: 1
Other: Placebo — placebo pill of the same size, color, and shape as the dietary supplement.
  Arms: 2

SUMMARY:
This study is being done to detect the metabolic changes that Omega 3 fatty acid treatment has on the brain and to find out whether magnetic resonance spectroscopy (MRS) scan can detect metabolic differences between bipolar patients and healthy control participants.

DETAILED DESCRIPTION:
Bipolar disorder (BP) is a chronic, complex and highly heterogeneous disease that has been unrecognized or misdiagnosed in prepubertal children and adolescents. It is one of the most disabling forms of childhood psychopathology and carries a striking human and economic cost. A high percentage of children and adolescents with BP respond very poorly to existing treatments. There is a significant need for studies identifying the developmentally sensitive targets for novel therapeutic compounds for this truly disabling illness. A growing range of novel therapeutic options for the treatment of BP are under investigation. Highly unsaturated fatty acids of the omega-3 fatty acids are among the novel therapeutic compounds considered in the treatment of adult patients with BP. However, the mood-stabilizing efficacy and the neurometabolic effects of this naturally occurring dietary components have not been examined in pediatric patients with BP.

The objective of this study is to identify magnetic resonance spectroscopic characteristics of adolescents with BP before and during a double-blind, placebo controlled combined omega-3 fatty and omega -6 fatty acid trial. We will compare the spectroscopic findings of the BP group with individually matched healthy comparison subjects before and after the omega-3/omega-6 fatty acid treatment. We will identify a well-described cohort of adolescents (age: 12-18) with BP without catatonic features, psychotic features, or other psychiatric comorbidity. Comorbidity with ADHD will be allowed since this might be a separate phenotype for pediatric BP. We will analyze the differences between BP subjects with comorbid ADHD, and BP subjects without ADHD. We will evaluate subjects with a novel magnetic resonance imaging technique, Magnetic Resonance Spectroscopic Imaging (MRSI). We will use a high-field 3T magnet to perform the MRSI acquisition, and apply a tissue volume correction technique to compare absolute metabolite concentrations rather than metabolite ratios. Previous studies found pronounced abnormalities in the frontal lobes, cingulate cortex, thalamus and basal ganglia of patients with BP. Thus, the region of interest in this study will include these anatomical areas with special emphasis given to prefrontal cortex and anterior cingulate cortex.

To our knowledge, this will be the first study examining omega-3 fatty acid induced changes in the developing brain in vivo. The long-term goal of our research group is to identify the developmentally sensitive, trait and state related magnetic resonance spectroscopic markers of pediatric BP. The preliminary data obtained from this application will be used to design a larger scale, follow-up study to examine whether alterations in brain metabolite measures are clinical state or trait markers and to determine the developmental variability in the patterns of metabolic abnormalities. Such knowledge will provide powerful insight into developmentally sensitive targeted pharmacological interventions. Studying bipolar disorder early in its course will be important to minimize potentially confounding factors, such as the effects of long-term medication use and neurodegeneration related to chronic illness course and substance abuse.

Based on the existing literature, we hypothesized that increased myoinositol levels will be detected in the regions of interests of adolescents with BP in comparison to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 18 years old
* both male and female
* all ethnic backgrounds
* DSM-IV criteria for Bipolar Disorder without catatonic and psychotic features or other psychiatric comorbidity, except ADHD

Exclusion Criteria:

* cardiac pacemakers
* metallic clips
* other bodily metallic implants
* dental braces
* not fluent in English

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Cases will classify as either treatment responders or non. Using dichotomous assessment, logistic regression will assess association of regional mI levels and mood measures taken at baseline, adjusting for important covariates such as age and gender. | at the 12 week point

CONTACTS AND LOCATIONS:
Overall Officials: Sencan S Unal, M.D. P, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States